CLINICAL TRIAL: NCT01703039
Title: Riluzole Augmentation Pilot in Depression (RAPID) Trial
Acronym: RAPID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI departure, slow recruitment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Harder, Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012P001841
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depression; Major Depressive Disorder; Depression; Riluzole; Glutamate; Sertraline
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Riluzole; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sertraline + riluzole (Experimental): sertraline 100 mg po daily and riluzole 50 mg po bid
  Interventions: Drug: Riluzole; Drug: Sertraline
- sertraline + placebo (Active Comparator): sertraline 100 mg po daily and placebo
  Interventions: Drug: Sertraline; Other: placebo

INTERVENTIONS:
Drug: Riluzole
  Other Names: Rilutek
  Arms: sertraline + riluzole
Drug: Sertraline
  Other Names: Zoloft
Other: placebo
  Arms: sertraline + placebo

SUMMARY:
The investigators are doing a research study to find out if riluzole, when taken along with a standard antidepressant (sertraline) can help people with major depression.

This research study will compare riluzole + sertraline to placebo + sertraline. The investigators hypothesize that adding riluzole will lead to a better antidepressant response, in less time, then sertraline alone.

DETAILED DESCRIPTION:
Recent attention has focused on the glutamatergic system as a new, distinct target for depression treatment. Riluzole (Rilutek, Sanofi), an oral modulator of glutamate activity with neuroprotective and anticonvulsant properties, is currently approved by the United States Food and Drug Administration for treatment of amyotrophic lateral sclerosis (ALS). Preliminary studies using riluzole to treat depression in humans are promising, though larger, double-blinded controlled trials are needed.

Overall study population:

Adult outpatients with a current, untreated major depressive episode.

Disallowed therapies include: other psychotropic medications, including antipsychotics, mood stabilizers, benzodiazepines, barbiturates, other sedative-hypnotics, chronic opiates, or additional antidepressants, psychotherapy, electroconvulsive therapy, vagal nerve stimulations therapy, transcranial magnetic stimulation therapy, or phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18-75) who meet DSM-IV criteria for a major depressive episode,
* Hamilton Depression Rating Scale (HDRS) >22, and
* No antidepressant treatment for at least three weeks

Exclusion Criteria:

* Active drug or alcohol disorder in the past 3 months
* History of psychosis, history of mania or hypomania
* Epilepsy or history of seizures
* Hypothyroidism
* Congenital QTc prolongation
* Liver disease
* Lung disease
* Acute suicide or homicide risk
* Pregnant women, breastfeeding women, women of childbearing age not using contraception
* Unstable medical illness
* Elevated thyroid-stimulating hormone (TSH>5.0mlU/L), or
* Abnormal liver function tests (ALT>50 U/L or AST>50 U/L)
* ADD / ADHD (Attention deficit hyperactivity disorder)

Disallowed therapies include: other psychotropic medications, including antipsychotics, mood stabilizers, benzodiazepines, barbiturates, other sedative-hypnotics, chronic opiates, or additional antidepressants, psychotherapy, electroconvulsive therapy, vagal nerve stimulations therapy, transcranial magnetic stimulation therapy, or phototherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Harder, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline + Riluzole: sertraline 100 mg po daily and riluzole 50 mg po bid
  Riluzole
  Sertraline
- Sertraline + Placebo: sertraline 100 mg po daily and placebo
  Sertraline
  placebo
Period: Overall Study
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo
Started | 9 | 12
Completed | 6 | 7
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.83 (14.88) | 52.86 (7.71) | 53.31 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 13
Hamilton Depression Rating Scale (HDRS) [Mean (Standard Deviation); unit: units on a scale] — Scale measures presence and severity of depression. Scale ranges from a minimum score of 0 to a maximum score of 52. Higher values represent more severe depression and a worse outcome.
  units on a scale | 26 (2.53) | 25.14 (2.97) | 25.54 (2.70)
Hamilton Anxiety Rating Scale (HARS) [Mean (Standard Deviation); unit: units on a scale] — Scale measures anxiety. Total highest score is 56. Higher scores indicate worse anxiety.
  units on a scale | 29.83 (7.33) | 27.14 (10.12) | 28.38 (8.69)
Clinical Global Impression Scale (CGI) [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression (CGI) severity of illness scale rates overall severity of illness.
  CGI scores range from 1 to 7. Higher scores are worse outcomes.
  units on a scale | 5 (0.63) | 5.14 (0.90) | 5.08 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hamilton Depression Rating Scale (HDRS) Score From Baseline (0 Weeks) to Endpoint at 8 Weeks
Description: The Hamilton Depression Rating Scale (HDRS) is a clinician-administered semi-structured interview with 17 questions. It is designed to measure the severity of depressive symptoms in patients with a primary depressive illness. Higher HDRS scores indicate a worse outcome. The scale has a minimum value of 0 and a maximum value of 52.
Time Frame: 0 weeks-8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sertraline + Riluzole: sert 100mg po daily and riluzole...
- Sertraline + Placebo: sert 100mg po daily and placebo...
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo
Number analyzed (Participants) | 6 | 7
score on a scale | -5.67 (7.09) | -13.43 (6.53)
Statistical Analysis 1: Comparison: Sertraline + Riluzole vs Sertraline + Placebo; Test type: Superiority; p = 0.06, ANOVA

2. Primary Outcome: Number of Patients Experiencing an Antidepressant Response (>50% Reduction in HDRS) at Endpoint of 8 Weeks
Description: as for outcome 1
Time Frame: 0 weeks-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo
Number analyzed (Participants) | 6 | 7
Participants | 1 | 3
Statistical Analysis 1: Comparison: Sertraline + Riluzole vs Sertraline + Placebo; Test type: Superiority; p = 0.31, Chi-squared

3. Primary Outcome: Number of Patients Experiencing Remission From Depression (HDRS<7) at Endpoint of 8 Weeks
Description: as for outcome 1
Time Frame: 0 weeks-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo
Number analyzed (Participants) | 6 | 7
Participants | 0 | 1
Statistical Analysis 1: Comparison: Sertraline + Riluzole vs Sertraline + Placebo; Test type: Superiority; p = 0.34, Chi-squared

4. Secondary Outcome: Mean Change in Hamilton Anxiety Rating Scale (HARS) Score From Baseline (0 Weeks) to Endpoint at 8 Weeks
Description: The HARS scale is a clinician rated interview scale designed to measure the signs and symptoms of anxiety. It has 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) were summed up to give a total possible score of 0 (not present) to 56 (very severe), where lower scores indicate less anxiety.
Time Frame: 0 weeks-8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo
Number analyzed (Participants) | 6 | 7
score on a scale | -9.50 (10.88) | -15.57 (7.72)
Statistical Analysis 1: Comparison: Sertraline + Riluzole vs Sertraline + Placebo; Test type: Superiority; p = 0.27, ANOVA

5. Secondary Outcome: Mean Change in Clinical Global Impression (CGI) Scale From Baseline (0 Weeks) to Endpoint at 8 Weeks
Description: The Clinical Global Impression Scale (CGI) is a brief clinician-rated instrument. The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Treatment response ratings should take account of both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side-effects) and 4 (unchanged or worse and side-effects outweigh the therapeutic effects). Each component of the CGI is rated separately; the instrument does not yield a global score.
Time Frame: 0 weeks-8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo
Number analyzed (Participants) | 6 | 7
score on a scale | -0.67 (0.82) | -2.71 (1.98)
Statistical Analysis 1: Comparison: Sertraline + Riluzole vs Sertraline + Placebo; Test type: Superiority; p = 0.04, ANOVA

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Sertraline + Riluzole | Sertraline + Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 2/9 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline + Riluzole (N=9) | Sertraline + Placebo (N=12)
Nausea (Gastrointestinal disorders) | 1 | 0
Elevated Liver Function Tests (LFTs) (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT01703039/Prot_SAP_000.pdf